CLINICAL TRIAL: NCT03828227
Title: Phase III Study to Evaluate the Quality of Life in Elderly Patients With Metastatic Colorectal Cancer Receiving First-line Therapy Based on Simplified Geriatric Parameters.
Brief Title: QoL in mCRC Elderly Patients Receiving First-line Therapy Based on Simplified Geriatric Parameters.
Acronym: COLAGE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COLAGE C18-01 PRODIGE 66
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Elderly Patients; Metastatic Colorectal Cancer; Quality of Life
Keywords: chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Candidate group" OPTIMOX plus bevacizumab (Arm A) (Active Comparator): Patients with :
  * Serum albumin level ≥ 30g/L,
  * ECOG PS 0-1 (whatever mini GDS score) or ECOG PS 2 with mini GDS 0 (ie, no depression).
  Adapted FOLFOX7 (aFOLFOX7)-bevacizumab for 6 cycles and then Adapted LV5FU2 (aLV5FU2)-bevacizumab (until progression or or unacceptable limiting toxicity)
  Interventions: Drug: OPTIMOX-bevacizumab
- "Candidate group" - Capecitabine-bevacizumab (Arm B) (Active Comparator): Patients with :
  * Serum albumin level ≥ 30g/L,
  * ECOG PS 0-1 (whatever mini GDS score) or ECOG PS 2 with mini GDS 0 (ie, no depression).
  This treatment regimen will be given until disease progression (PD) or unacceptable limiting toxicity, as follows:
  Interventions: Drug: Capecitabine plus bevacizumab
- "Non candidate group" - Capecitabine-bevacizumab (Active Comparator): Patients with:
  * Serum albumin level < 30g/L.
  * And/ or ECOG PS 2 and mini GDS ≥ 1 (ie, depression).
  This treatment regimen will be given until disease progression (PD) or unacceptable limiting toxicity, as follows:
  Interventions: Drug: Capecitabine plus bevacizumab

INTERVENTIONS:
Drug: OPTIMOX-bevacizumab — Induction Adapted FOLFOX7 (aFOLFOX7)-bevacizumab for 6 cycles (3 months)
  * Bevacizumab: 5 mg/kg IV (day 1, every 2 weeks [q2w]),
  * Folinic acid (FA): 400 mg/m² IV/2h (day 1, q2w),
  * Oxaliplatin: 85 mg/m² IV/2h (day 1, q2w),
  * 5-fluorouracil (5-FU) continuous infusion 2400 mg/m² IV/46h (day 1-2, q2w),
  * No 5-FU bolus.
  then Maintenance Adapted LV5FU2 (aLV5FU2)-bevacizumab (until progression or or unacceptable limiting toxicity)
  * Bevacizumab: 5 mg/kg IV (day 1, q2w),
  * FA: 400 mg/m² IV/2h (day 1, q2w),
  * 5-FU continuous infusion 2400 mg/m² IV/46h (day 1-2, q2w)
  * No 5-FU bolus
  Other Names: Folinic acid (FA)-5-fluorouracil (5-FU)-oxaliplatin [OPTIMOX]; Avastin
  Arms: "Candidate group" OPTIMOX plus bevacizumab (Arm A)
Drug: Capecitabine plus bevacizumab — * Bevacizumab: 7.5 mg/kg intravenous infusion [IV] (day 1; q3w),
  * Capecitabine: 1000 mg/m² orally twice a day (day 1 through day 14, q3w).
  Other Names: capecitabine; Avastin
  Arms: "Candidate group" - Capecitabine-bevacizumab (Arm B); "Non candidate group" - Capecitabine-bevacizumab

SUMMARY:
A national, multicenter, open-label, randomized phase III study. The trial aim is to determine the best therapeutic strategies according with the HRQoL.

DETAILED DESCRIPTION:
Treatment cohort will be determined based on three parameters:

* Serum albumin level at baseline,
* ECOG Performance Status,
* Mini GDS.

The "Candidate" group will be defined according to (all the following criteria must be fulfilled):

* Serum albumin level ≥ 30g/L,
* ECOG PS 0-1 (whatever mini GDS score) or ECOG PS 2 with mini GDS 0 (ie, no depression).

The "Non-candidate" cohort group will be defined according to (at least one of those parameters is fulfilled):

* Serum albumin level < 30g/L.
* And/ or ECOG PS 2 and mini GDS ≥ 1 (ie, depression).

Patients in the "Candidate group" will be randomized to:

* OPTIMOX bevacizumab (arm A),
* Capecitabine + bevacizumab (arm B), in priority followed by FOLFOX-bevacizumab at first progression.

Patients in the "Non-candidate" group cohort

- Not randomized, follow-up patients receiving: capecitabine + bevacizumab

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically proven colorectal adenocarcinoma,
3. Confirmed metastatic disease,
4. Patients with no detected dihydropyridine dehydrogenase (DPD) deficiency,
5. No prior therapy for metastatic disease (in case of previous adjuvant chemotherapy, interval between the end of chemotherapy and relapse must be > 6 months for fluoropyrimidine alone or > 12 months for oxaliplatin-based chemotherapy,
6. Duly documented unresectable metastatic disease i.e., not suitable for complete carcinological surgical resection,
7. Age ≥ 75 years,
8. ECOG PS 0-2,
9. Hematological status: neutrophils ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, and hemoglobin > 9 g/dL,
10. Adequate renal function: serum creatinine level < 150 µmol/l, and creatinine clearance (Cockcroft and Gault or MDRD formula > 30 mL/min),
11. Adequate liver function: total bilirubin level < 1.5 x upper normal limit (ULN), serum alkaline phosphatase (ALP) level < 5 x ULN,
12. Proteinuria < 2+ (dipstick urinalysis) or ≤ 1g/24h,
13. Regular follow-up feasible. The registered patient must be treated and followed at the participating center,
14. Registration in France with the French National Health Care System (including dispositive PUMA (protection Universelle Maladie).

Exclusion Criteria:

1. History or evidence upon physical examination of CNS metastasis (e.g. non- irradiated CNS metastasis, seizure not controlled with standard medical therapy), unless adequately treated,
2. Neuropathy grade > 1,
3. Patient with known dihydropyridine dehydrogenase (DPD) deficiency or history of severe and unexpected reactions to a fluoropyrimidine-containing regimen, or in case of clinically significant active heart disease or myocardial infarction within 6 months or if patient treated with sorivudine or its clinically related analogues, such as brivudine
4. Uncontrolled hypercalcemia,
5. Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy,
6. Medical history of other concomitant or previous malignant disease, except adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer in complete remission for ≥ 5 years,
7. History of arterial thrombotic and/or embolic event (e.g. myocardial infarction, stroke…) within 6 months prior to randomization,
8. History of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to randomization,
9. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding,
10. Major surgery (open biopsy, surgical resection, wound revision or any other major surgery involving entry into body cavity) or significant traumatic injury within the last 28 days prior to randomization, and/or minor surgical procedure including placement of a vascular device within 2 days of first study treatment,
11. Concomitant administration of prophylactic phenytoin,
12. Treatment with sorivudine or its chemically related analogues, such as brivudine,
13. Patients with known allergy/hypersensitivity to any component of study drugs
14. Concomitant unplanned anti-tumor treatment,
15. Participation in another clinical trial with any investigational drug within 30 days prior to randomization,
16. Other serious and uncontrolled non-malignant disease,
17. Patient under guardianship, curatorship or under the protection of justice

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) at 6 months in the "candidate group". | At 6 months
  Improvement of HRQoL at 6 months by 10 points compared to the score at inclusion on the following targeted dimensions: emotional functioning (4 items) and global health (2 items) (score from 6-30 with higher values representing better quality of life).

SECONDARY OUTCOMES:
Number of patients amenable to second-line therapy. | until 58 months
  Proportion of patients amenable to second-line therapy.
Number of patient amenable to surgery and/or locoregional therapy. | until 58 months
  Proportion of patients amenable to salvage surgery and/or locoregional therapy (e.g., radiofrequency ablation, stereotactic radiotherapy, …).
Progression-free survival (PFS) | until 58 months
  PFS is defined as time from date of first dose of study treatment to date of first documented PD or death due to any cause determined by the Investigator assessment in accordance to RECIST 1.1. Alive patients without progression will be censored at the last tumor assessment, either during study treatment period or during follow-up period.
Overall survival (OS) | Until 58 months
  OS defined as the time between the date of the first dose of study treatment and the death date. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period.
Other dimensions of health-related quality of life (HRQoL) and longitudinal HRQoL | Until 58 months
  HRQoL: all other dimensions of the QLQC-30 and QLQELD-14 questionnaires, and longitudinal analyses of the QLQC-30 and QLQELD-14 elderly specific module integrating all measurement times.
Determination of instrumental activities of daily living (IADL) as prognostic factor for overall survival (OS). | Until 58 months
  IADL as prognostic factor for overall survival (OS) and treatment toxicity.
G8 score at baseline. | until 58 months
  To determine G8 score at baseline and to correlate the candidate group and the non-candidate group according to G8 score.
Performance status geriatric (PSG) score. | until 58 months
  External analysis of PSG score as predictive for treatment efficacy: PFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth CAROLA, MD, Principal Investigator — UCOG Picardie Groupe Hospitalier Public du Sud de l'Oise (GHPSO)
Locations (22):
- France (22):
  - CH Abbeville, Abbeville
  - CHU Amiens Hôpital sud, Amiens
  - Clinique de l'Europe, Amiens
  - CH Beauvais, Beauvais
  - Hôpital Duchenne, Boulogne-sur-Mer
  - Centre hospitalier de Cannes, Cannes
  - CH Compiègne Noyon, Compiègne
  - UCOG Picardie Groupe Hospitalier, Creil
  - CHU Henri Mondor, Créteil
  - Centre geroges François Leclerc, Dijon
  - Institut Daniel Hollard, Grenoble
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CH Sud Ile de France, Melun
  - CH Mont de Marsan, Mont-de-Marsan
  - Centre Antoine Lacassagne, Nice
  - Hôpital des Diaconnesses Croix Saint Simon, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CH Annecy Genevois, Pringy
  - CH Saint Malo, St-Malo

IPD SHARING:
Plan to Share IPD: No